CLINICAL TRIAL: NCT05935956
Title: An Observational, Single Arm, Open Label Study Evaluating the Safety and Effectiveness of Magnetic Peripheral Nerve Stimulation (mPNS) for the Treatment of Chemotherapy Induced Neuropathy (mPNS-CH)
Brief Title: Safety and Effectiveness of Magnetic Peripheral Nerve Stimulation for the Treatment of Chemotherapy Induced Neuropathy
Acronym: mPNS-CH
Status: Completed | Type: Observational
Sponsor: NeuraLace Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NLM-005
Record Dates: First submitted 2023-06-12; First posted 2023-07-07 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2023-07

CONDITIONS: Neuralgia; Neuropathic Pain; Chemotherapy-induced Peripheral Neuropathy
Keywords: Transcutaneous Magnetic Peripheral Nerve Stimulation; Axon Therapy; Peripheral Neuropathy; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: conditions — Neuralgia; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Magnetic Peripheral Nerve Stimulation — Magnetic Peripheral Nerve Stimulation
  Other Names: Axon Therapy

SUMMARY:
Assess the safety and effectiveness of Axon Therapy in the treatment of chemotherapy-induced neuropathy

DETAILED DESCRIPTION:
This is an observational, single arm, open label study in which up to 20 subjects diagnosed with chemotherapy induced neuropathy will be treated with mPNS.

Subjects will be consented, screened, and undergo a 7-day baseline assessment to measure pain scores and assess diary compliance. Subjects who meet inclusion criteria will undergo an in-clinic baseline evaluation and start their treatment.

All subjects will return to the clinic for follow-up assessment at Day 30 (± 14 days) and Day 90 (± 14 days) and will return to the clinic for mPNS treatments as follows:

* Month 1: 6 treatments

  * WEEK 1: 3 treatments (consecutive treatments are best)
  * WEEK 2-4: Weekly treatments
* Month 2: Bi-Weekly treatment
* Month 3: Treatments every 2-4 weeks
* Additional treatments to treat flare ups; defined as an episode of pain with a VAS of at least 5 following an increase in daily activities.
* The Lead Investigator is provided the discretion to modify the treatment protocol based on subject response.

In addition to in-clinic assessments and treatments, all subjects will complete an electronic twice daily diary through 90 days of the study. Subjects will receive weekly phone follow-up for diary reminders and to assess for the occurrence of adverse events after treatment starts. Weekly phone follow-ups will only occur during weeks when the subject is not seen in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the study.
2. Subject is willing and able to comply with scheduled visits, treatment plan, daily pain, and other study procedures subject is able and willing to complete twice daily diary for 90 days.
3. Subject must be literate in English to fill out the study questionnaires.
4. Men or women of any race or ethnicity who are 18-85 years of age.
5. Subject must have chemotherapy induced neuropathy for more than three months per medical history.
6. Subject has a pain score >5 on a VAS at Enrollment/Screening Visit.
7. Subject has completed at least one of the two daily pain diary entries on at least three days between the Enrollment/Screening Visit and Visit 1 with a mean pain score of ≥4 and <10 based on Daily VAS to be eligible for the study.
8. Subject has been on a stable pain medication regimen for at least 28 days, as determined by the investigator or is not taking pain medications, at the baseline assessment in this study.

Exclusion Criteria:

1. Subjects with neuropathic pain due to post-herpetic neuropathy, HIV, trigeminal neuralgia, carpal or tarsal tunnel syndrome; subjects whose post-traumatic neuropathic pain is categorized as central (e.g., spinal cord injury) rather than peripheral.
2. Subject has a currently diagnosed progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, or severe/critical spinal stenosis (stenosis).
3. Subjects with skin conditions in the affected dermatome that in the judgment of the investigator could interfere with evaluation of the neuropathic pain condition.
4. Subjects with other pain that may confound assessment or self-evaluation of the peripheral neuropathic pain.
5. Participation in any other clinical trial within 30 days prior to screening and/or during participation in this study.
6. Any subject considered at risk of suicide or self-harm based on investigator judgment and/or the details of a risk assessment.
7. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality, or other factors that may increase the risk associated with study participation or investigational product administration or may interfere with compliance or the interpretation of study results and, in the judgment of the investigator would make the subject inappropriate to participate in the study.
8. Subjects with pending Worker's Compensation, civil litigation, or disability claims; Subjects with fully resolved litigation and compensation claims can participate.
9. Phantom limb pain or pain that feels like it is coming from a body part that is no longer there.
10. Subjects with shrapnel or ferromagnetic objects
11. Subject is currently taking a morphine equivalent daily dose > 120 mg/day.
12. Subject is currently pregnant or is a woman of childbearing potential, not using adequate contraception or not willing to comply with contraception for the duration of the study.
13. Subjects with active drug or alcohol abuse within 1 year prior to screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately twenty (20) subjects aged 18-85 years old and presenting with chemotherapy induced neuropathy will be enrolled at 1 site in the United States.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Effectiveness of mPNS for treating chemotherapy-induced neuropathy, measured by a reduction in pain at Day 90 as compared to Baseline, using a visual analog scale (VAS). | 90 days
  The primary effectiveness endpoint is to demonstrate a reduction in pain at Day 90 as compared to Baseline where pain is measured in-clinic using a visual analog scale (VAS). Scores on the VAS range from 0 (no pain) to 10 (worst possible pain).
Safety of mPNS for the treatment of chemotherapy-induced neuropathy, as measured by the incidence of therapy-related adverse events (AEs) through Day 90. | 90 days
  The primary safety endpoint is the occurrence of therapy-related adverse events (AEs) through Day 90.

SECONDARY OUTCOMES:
Patient Reported Outcome (PRO) assessment via the Pain Disability Index (PDI), which measures the degree that chronic pain interferes with normal role functioning. | Baseline and 90 days
  The PDI is a short, self-reported instrument for measuring the degree of interference with normal role functioning caused by chronic pain. The form uses a 10-point scale ranging from 0 (no disability) to 10 (total disability) to rate pain-related interference in the following categories: family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity. The total scores range from a minimum of 0 to a maximum of 70, where a higher score indicates higher pain-related interference.
PRO assessment via the EuroQol Group Quality of Life Questionnaire (EQ-5D-3L), which measures the impact that chronic pain has on 5 aspects of a subject's quality of life. | Baseline and 90 days
  The EQ-5D-3L is a descriptive questionnaire comprised of 5 dimensions; each describing a different aspect of health: Mobility; Self-Care; Usual Activities; Pain/Discomfort and Anxiety/Depression on a 3-level response scale. The three levels represent no problem, some/moderate problems, and severe/extreme problems across the 5 dimensions. The EQ-5D-3L summary index is derived by combining one level from each of the 5 dimensions and converting it to a single summary index or health utility value, which ranges from 0 for worst imaginable health state to 100 for best imaginable health state. Together 243 health states are possible (35 combinations). Overall scores for the EQ-5D-3L index range from -0.109 to 1, with low scores representing a higher level of dysfunction and hence, a worse outcome.
PRO assessment via the Daily Sleep Interference Scale (DSIS), which measures how much a subject's pain interferes with that subject's sleep. | Baseline and 90 days
  The DSIS describes the degree that pain has interfered with the subject's sleep. Response options range from 0 (Did not interfere with sleep) to 10 (Completely interfered with sleep-unable to sleep due to pain). A lower score indicates a better outcome.
PRO assessment via the Depression Anxiety Stress Scales (DASS), which measures the level of depression, anxiety and stress a subject is experiencing. | Baseline and 90 days
  The DASS is a 42-item, self-reported rating inventory that measures depression, anxiety, and stress. Each answer is scored on a scale of 0-3 with a total minimum score of 0 and maximum of 126. Scores from 0-9 indicate a normal score, scores of 10-13 indicate mild depression, scores of 14-20 indicate moderate depression, scores of 21-27 indicate severe depression and scores, and a score greater than 28 indicates extremely severe depression.
PRO assessment via the Brief Pain Inventory (BPI-SF) to assess the severity of pain and the impact of pain on daily functions. | Baseline and 90 days
  The BPI-SF is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions. The BPI-SF consists of 5 questions. Four items measure pain on 11-point response scales from 0 to 10 ("No Pain" to "Pain as bad as you can imagine"). Another item, containing 7 sub-questions, evaluates the level of pain interference with daily functioning on 11-point response scales from 0 to 10 ("Does not interfere" to "Completely interferes"). Lower scores indicate better outcomes.
PRO assessment via the Patient Global Impression of Change (PGIC), which measures patient satisfaction after treatment with magnetic peripheral nerve stimulation (NeuraLace Axon Therapy) | Day 90
  The PGIC is a self-administered instrument that measures the proportion of subjects in each PGIC satisfaction category that has improved post-treatment with magnetic peripheral nerve stimulation (NeuraLace Axon Therapy), based on a scale ranging from 1 (very much improved) to 7 (very much worse). The subject is presented with a 7-point rating scale containing the options "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", and "very much worse". A lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Johnson, MD, PhD, Principal Investigator — Carolinas Pain Institute and Center for Clinical Research
Locations (1):
- Carolinas Pain Institute and Center for Clinical Research, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No